CLINICAL TRIAL: NCT01496313
Title: An International, Randomised, Double-Blind, Two-Arm Study To Evaluate The Safety And Efficacy Of Vandetanib 150 And 300mg/Day In Patients With Unresectable Locally Advanced Or Metastatic Medullary Thyroid Carcinoma With Progressive Or Symptomatic Disease
Brief Title: To Compare The Effects Of Two Doses Of Vandetanib In Patients With Advanced Medullary Thyroid Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D4200C00097; LPS14809 (Other: Sanofi Identifier); 2011-004701-24 (EudraCT Number)
Record Dates: First submitted 2011-12-02; First posted 2011-12-21 (Estimated); Results first posted 2015-11-27 (Estimated); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Thyroid Cancer
Keywords: medullary thyroid cancer; metastatic; thyroid cancer; carcinoma of the thyroid; receptor tyrosine kinase inhibitor; VEGFR; Unresectable locally advanced thyroid cancer
MeSH Terms: conditions — Thyroid Neoplasms; Carcinoma, Medullary; Neoplasm Metastasis | interventions — vandetanib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- 300mg vandetanib (Active Comparator)
  Interventions: Drug: 300mg vandetanib
- 150mg vandetanib (Active Comparator)
  Interventions: Drug: 150mg vandetanib

INTERVENTIONS:
Drug: 300mg vandetanib — Oral blinded tablets taken once daily.
  At objective disease progression or 14 months (whichever is earlier), patient may be unblinded to treatment
  Dosing with unblinded study treatment can continue until 24 months after patient was randomised.
  At any time dosing may be interrupted for up to 6 weeks due to toxicity. Dosing may restart at a reduced dose (200mg/day). Once reduced, dose increases are not permitted and dosing must stop if further toxicities occur.
  Other Names: SAR390530
  Arms: 300mg vandetanib
Drug: 150mg vandetanib — Oral blinded tablets taken once daily.
  At objective disease progression or 14 months (whichever is earlier), patient may be unblinded to treatment. Patients who have not dose reduced at the time of unblinding may have their dose increased to 300mg
  Dosing with unblinded study treatment can continue until 24 months after patient was randomised
  At any time dosing may be interrupted for up to 6 weeks due to toxicity. Dosing may restart at a reduced dose (100mg/day) [OR 300 reduced to 200mg/day if dose was increased at unblinding.] Once reduced, dose increases are not permitted and dosing must stop if further toxicities occur.
  Other Names: SAR390530
  Arms: 150mg vandetanib

SUMMARY:
The purpose of this study is to give patients with medullary thyroid cancer either 300mg/day or 150mg/day vandetanib and compare how well each dose affects how their cancer responds. It will also help the investigators understand the side effects of different doses in these patients.

DETAILED DESCRIPTION:
An International, Randomised, Double-Blind, Two-Arm Study To Evaluate The Safety And Efficacy Of Vandetanib 150 And 300mg/Day In Patients With Unresectable Locally Advanced Or Metastatic Medullary Thyroid Carcinoma With Progressive Or Symptomatic Disease

ELIGIBILITY:
Inclusion Criteria:

* Written consent from Female or male patients aged 18 years and over. Previously confirmed histological diagnosis of unresectable, locally advanced or metastatic, hereditary or sporadic MTC Objective disease progression within the previous 14 months prior to enrolment, and/or
* Have one or more symptoms that the Investigator believes to be related to the patient's MTC.
* World Health Organisation (WHO) or Eastern Cooperative Oncology Group (ECOG) Performance status 0-2.
* Has measurable disease (at least one lesion, not irradiated within 12 weeks of study randomisation, with longest diameter more or equal 10mm (lymph nodes minimum more or equal 15 mm) with CT or MRI).
* Lesions must be amenable to accurate and repeat measurement.

Exclusion Criteria:

* Prior treatment (major surgery, radiation therapy, chemotherapy, or other investigational drugs) received within 28 days before randomization.
* Abnormal liver function tests (bilirubin more than 1.5xULRR, and ALT, AST, or ALP more than 2.5xULRR or 5.0xULRR if related to liver metastases).
* Significant cardiac conditions or events such as reduced cardiac functions, symptomatic cardiac arrhythmia requiring treatment, congenital long QT syndrome, history of drug-induced QT prolongation, or QTcF correction unmeasurable or more than 450 ms.
* Abnormal electrolytes such as potassium, magnesium and calcium, or abnormal organ functions such as decreased creatinine clearance.
* For women only - currently pregnant or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2012-06-08 (Actual); Primary Completion 2014-04-02 (Actual); Study Completion 2024-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Chair — Sanofi
Locations (30):
- Research Site, Houston, Texas, United States
- Czechia (4):
  - Investigational Site Number : 1903, Olomouc
  - Research Site, Olomouc
  - Investigational Site Number : 1901, Prague
  - Research Site, Prague
- India (2):
  - Research Site, Bangalore Karnataka
  - Research Site, Vellore
- Israel (4):
  - Research Site, Beersheba
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Petah Tikva
- Italy (7):
  - Research Site, Catania
  - Research Site, Milan
  - Research Site, Palermo
  - Research Site, Pisa
  - Research Site, Roma
  - Research Site, Siena
  - Research Site, Torino
- Netherlands (2):
  - Research Site, Groningen
  - Research Site, Leiden
- Poland (5):
  - Investigational Site Number : 5704, Warsaw, Masovian Voivodeship
  - Investigational Site Number : 5703, Gliwice
  - Research Site, Gliwice
  - Research Site, Warsaw
  - Research Site, Zgierz
- Research Site, Saint Petersburg, Russia
- United Kingdom (4):
  - Research Site, Cardiff
  - Research Site, Greater London
  - Research Site, London
  - Research Site, Tyne & Wear

REFERENCES:
- See also: D4200C00097_CSR_Synopsis.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1434&filename=D4200C00097_Study_Synopsis.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 8 June 2012 to 2 April 2014, 81 participants were randomized by 29 centers in 9 global countries. The study consisted of a double-blind randomized period and an open-label period.
Pre-assignment Details: 93 participants were screened; 81 participants were randomized to treatment. Participants with objective disease progression within the 14 months on blinded treatment were given the option to continue to receive vandetanib in open-label period for up to 2 years from the time of study entry. Participants were followed for efficacy during the randomized period only. No further efficacy data was collected in open-label period as pre-specified in the protocol.
Groups:
- Randomized Period: Vandetanib 150 mg; Randomized Period: Vandetanib 300 mg: Oral blinded tablet, taken once daily
- Open-label Period: Vandetanib 100 mg: Participants who received vandetanib 150 milligrams (mg) orally once daily but the dose was reduced to vandetanib 100 mg orally once daily for an adverse event (AE) or QT prolongation in randomized period continued receiving the reduced dose of vandetanib 100 mg orally once daily in open-label period as per the Investigator for a maximum of 2 years from study entry.
- Open-label Period: Vandetanib 150 mg: Participants who received vandetanib 150 mg orally once daily without any dose reduction for an AE or QT prolongation in randomized period were given an option to stay on vandetanib 150 mg orally once daily in open-label period for a maximum of 2 years from study entry.
- Open-label Period: Vandetanib 200 mg: Participants who received vandetanib 300 mg orally once daily but the dose was reduced to vandetanib 200 mg orally once daily for an AE or QT prolongation in randomized period continued receiving the reduced dose of vandetanib 200 mg orally once daily in open-label period as per the Investigator for a maximum of 2 years from study entry.
- Open-label Period: Vandetanib 300 mg: Participants who received vandetanib 150 mg or 300 mg orally once daily without any dose reduction for an AE or QT prolongation in randomized period were given an option to increase or continue vandetanib 300 mg orally once daily in open-label period respectively for a maximum of 2 years from study entry.
Period: Randomized Period (up to 14 Months)
Arm/Group | Randomized Period: Vandetanib 150 mg | Randomized Period: Vandetanib 300 mg | Open-label Period: Vandetanib 100 mg | Open-label Period: Vandetanib 150 mg | Open-label Period: Vandetanib 200 mg | Open-label Period: Vandetanib 300 mg
Started | 40 | 41 | 0 | 0 | 0 | 0
Completed (Completed treatment) | 35 | 26 | 0 | 0 | 0 | 0
Not Completed | 5 | 15 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 5 | 0 | 0 | 0 | 0
Not completed — Condition Under Investigation Worsened | 2 | 3 | 0 | 0 | 0 | 0
Not completed — Study-specific Discontinuation Criteria | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Participant Decision | 1 | 3 | 0 | 0 | 0 | 0
Not completed — Other | 1 | 2 | 0 | 0 | 0 | 0
Period: Open-Label Period (Month 14 to 2 Years)
Arm/Group | Randomized Period: Vandetanib 150 mg | Randomized Period: Vandetanib 300 mg | Open-label Period: Vandetanib 100 mg | Open-label Period: Vandetanib 150 mg | Open-label Period: Vandetanib 200 mg | Open-label Period: Vandetanib 300 mg
Started (Started open-label period) | 0 | 0 | 5 | 9 | 8 | 39
Completed | 0 | 0 | 3 | 7 | 7 | 28
Not Completed | 0 | 0 | 2 | 2 | 1 | 11
Not completed — Study-specific Withdrawal Criteria | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Participant Decision | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Other | 0 | 0 | 2 | 2 | 1 | 7

BASELINE CHARACTERISTICS:
Groups:
- Vandetanib 150 mg; Vandetanib 300 mg: Oral blinded tablet, taken once daily
- Total: Total of all reporting groups
Arm/Group | Vandetanib 150 mg | Vandetanib 300 mg | Total
Number analyzed (Participants) | 40 | 41 | 81
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.2 (15.24) | 52.7 (15.42) | 52.5 (15.24)
Age, Customized [Number; unit: Participants]
  >=18 to <40 years | 9 | 9 | 18
  >=40 to <65 years | 22 | 20 | 42
  >=65 to <75 years | 7 | 10 | 17
  >=75 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 12 | 27
  Male | 25 | 29 | 54
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 1 | 2 | 3
  Black or African American | 0 | 1 | 1
  White | 39 | 37 | 76
  Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) for Vandetanib 150 and 300mg With Responses Determined by the Investigator
Description: ORR=proportion of patients with a best response of complete or partial response as per Response Evaluation Criteria in Solid Tumors(RECIST)1.1
Time Frame: Randomisation to week 60 (maximum)
Population: Per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), disappearance of all target lesions; Partial response (PR), at least a 30% decrease in the sum of diameters of target lesions; ORR = CR + PR
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Vandetanib 150 mg | Vandetanib 300 mg
Number analyzed (Participants) | 40 | 41
Proportion of participants | 0.20 [0.105 to 0.348] | 0.29 [0.176 to 0.445]

2. Secondary Outcome: Best Objective Response
Time Frame: Randomisation to week 60 (maximum)
Population: Per RECIST v1.1 for target lesions: CR, disappearance of all target lesions; PR, at least a 30% decrease in the sum of diameters of target lesions; Progressive disease (PD), at least 20% increase in the sum of diameters of target lesions; Stable disease (SD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD
Measure: Number; unit: Participants
Arm/Group | Vandetanib 150 mg | Vandetanib 300 mg
Number analyzed (Participants) | 40 | 41
Participants
  Complete response | 0 | 1
  Partial response | 8 | 11
  Stable disease | 21 | 23
  Progressive disease | 9 | 2
  Non-evaluable | 2 | 4

3. Secondary Outcome: Duration of Objective Response (RECIST 1.1) by Treatment Arm
Time Frame: Randomization to Week 60 (maximum)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vandetanib 150 mg | Vandetanib 300 mg
Number analyzed (Participants) | 8 | 12
Months | 9.8 [2.8 to 11.2] | 8.4 [3.0 to 11.2]

4. Secondary Outcome: Time to Objective Response (RECIST 1.1) by Treatment Arm
Time Frame: Randomization to Week 60 (maximum)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vandetanib 150 mg | Vandetanib 300 mg
Number analyzed (Participants) | 8 | 12
Months | 4.2 [2.8 to 11.2] | 4.4 [2.8 to 11.1]

5. Secondary Outcome: Percentage Change From Baseline in Target Lesion Size (RECIST 1.1) by Treatment Arm
Time Frame: Randomization to Week 60 (maximum)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | Vandetanib 150 mg | Vandetanib 300 mg
Number analyzed (Participants) | 40 | 41
% change
  Week 12 | -3.8 (29.24) | -17.5 (18.24)
  Week 24 | -13.0 (19.51) | -24.9 (22.11)
  Week 36 | -16.7 (24.33) | -29.1 (22.96)
  Week 48 | -20.7 (23.56) | -30.6 (25.31)
  Follow-up RECIST assessment | -51.0 (0) | -11.4 (67.05)
  Disc. of blinded vandetanib | -11.9 (27.98) | -27.3 (29.58)

6. Secondary Outcome: Plasma Concentration of Vandetanib in the Bloodstream (Cmax) for Patients by Treatment Arm.
Time Frame: Week 3 to week 60 (maximum)
Population: All patients who received at least 1 dose of vandetanib and for whom quantifiable plasma concentration data were available.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Vandetanib 150 mg | Vandetanib 300 mg
Number analyzed (Participants) | 40 | 41
ng/ml
  Week 3 (Day 21) | 428.6 (140.71) | 786.2 (243.15)
  Week 8 (Day 56) | 510.5 (206.50) | 941.0 (249.4)
  Week 12 (Day 84) | 561.4 (215.66) | 969.9 (396.18)
  Week 24 (Day 168) | 549.7 (189.62) | 1017.7 (330.89)
  Discontinuation of blinded vandetanib | 536.8 (225.34) | 964.0 (357.30)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and all-cause mortality (deaths) were collected from randomization (Day 1) up to end of follow-up, approximately 12 years. Other (non-serious) AEs were reported from randomization (Day 1) up to Week 108 (final analysis visit), 2 years.
Description: Analysis was performed on the safety population which included all participants who received at least 1 dose of randomized study drug (vandetanib) and for whom any post-dose data were available.
Groups:
- Open-label Period: Vandetanib 100 mg: Participants who received vandetanib 150 mg orally once daily but the dose was reduced to vandetanib 100 mg orally once daily for an AE or QT prolongation in randomized period continued receiving the reduced dose of vandetanib 100 mg orally once daily in open-label period as per the Investigator for a maximum of 2 years from study entry.
Arm/Group | Randomized Period: Vandetanib 150 mg | Randomized Period: Vandetanib 300 mg | Open-label Period: Vandetanib 100 mg | Open-label Period: Vandetanib 150 mg | Open-label Period: Vandetanib 200 mg | Open-label Period: Vandetanib 300 mg
All-Cause Mortality (participants affected / at risk) | 1/40 | 6/41 | 0/5 | 0/9 | 1/8 | 10/39
Serious Adverse Events (participants affected / at risk) | 9/40 | 9/41 | 0/5 | 4/9 | 2/8 | 11/39
Other Adverse Events (participants affected / at risk) | 38/40 | 40/41 | 5/5 | 7/9 | 7/8 | 31/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized Period: Vandetanib 150 mg (N=40) | Randomized Period: Vandetanib 300 mg (N=41) | Open-label Period: Vandetanib 100 mg (N=5) | Open-label Period: Vandetanib 150 mg (N=9) | Open-label Period: Vandetanib 200 mg (N=8) | Open-label Period: Vandetanib 300 mg (N=39)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina Pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac Failure Acute (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Duodenal Ulcer Perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis Erosive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug Interaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General Physical Health Deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sudden Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bile Duct Stone (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis Acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neurocysticercosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia Aspiration (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post Procedural Fistula (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft Tissue Necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma Pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Benign Laryngeal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Miller Fisher Syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral Motor Neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal Cord Compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Calculus Ureteric (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Laryngeal Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngeal Obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngeal Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized Period: Vandetanib 150 mg (N=40) | Randomized Period: Vandetanib 300 mg (N=41) | Open-label Period: Vandetanib 100 mg (N=5) | Open-label Period: Vandetanib 150 mg (N=9) | Open-label Period: Vandetanib 200 mg (N=8) | Open-label Period: Vandetanib 300 mg (N=39)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus Tachycardia (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 3 (3) | 5 (6) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Corneal Opacity (Eye disorders) | 2 (2) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye Pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Keratopathy (Eye disorders) | 6 (6) | 14 (17) | 2 (3) | 2 (2) | 0 (0) | 6 (7)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Anal Fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 15 (17) | 18 (21) | 0 (0) | 1 (1) | 2 (3) | 7 (7)
Dry Mouth (Gastrointestinal disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (5) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Asthenia (General disorders) | 5 (6) | 7 (7) | 1 (1) | 1 (1) | 0 (0) | 8 (10)
Fatigue (General disorders) | 8 (8) | 7 (7) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema Peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower Respiratory Tract Infection Bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia Staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash Pustular (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vulval Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthropod Bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Corneal Abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 5 (5) | 7 (7) | 0 (0) | 1 (1) | 0 (0) | 6 (7)
Aspartate Aminotransferase Increased (Investigations) | 3 (3) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 6 (7)
Blood Alkaline Phosphatase Increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood Bilirubin Increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood Creatine Phosphokinase Increased (Investigations) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood Creatinine Increased (Investigations) | 5 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Blood Glucose Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Thyroid Stimulating Hormone Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Thyroid Stimulating Hormone Increased (Investigations) | 12 (12) | 9 (11) | 0 (0) | 0 (0) | 1 (1) | 5 (8)
Ejection Fraction Decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Electrocardiogram Qt Prolonged (Investigations) | 5 (5) | 14 (15) | 1 (1) | 0 (0) | 1 (1) | 7 (8)
Gamma-Glutamyltransferase Increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Platelet Count Decreased (Investigations) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Weight Decreased (Investigations) | 2 (2) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
White Blood Cell Count Decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 2 (2) | 7 (8) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 7 (8) | 10 (11) | 2 (3) | 0 (0) | 0 (0) | 8 (9)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (3) | 7 (8) | 2 (3) | 1 (1) | 1 (1) | 6 (8)
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 (5) | 6 (9) | 2 (2) | 0 (0) | 1 (2) | 5 (6)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Iron Deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metastases To Bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Disturbance In Attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Head Titubation (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
Neuropathy Peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Depressed Mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 4 (6) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Micturition Urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 6 (7) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Renal Pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Dysaesthesia Pharynx (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Lower Respiratory Tract Inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 6 (7) | 6 (8) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 5 (5) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (4) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 8 (9) | 13 (19) | 0 (0) | 0 (0) | 1 (2) | 5 (5)
Rash Erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Cataract Operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 8 (10) | 11 (14) | 1 (1) | 1 (1) | 0 (0) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.